CLINICAL TRIAL: NCT03208725
Title: Building the Evidence Base for Appropriate Care of the Sick, Undernourished Child in Limited Resource Settings
Brief Title: Childhood Acute Illness and Nutrition Network
Acronym: CHAIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Washington (Other); Kenya Medical Research Institute (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); Makerere University (Other); Oregon Health and Science University (Other); The Hospital for Sick Children (Other); University of Amsterdam (Other); University of Malawi (Other); Aga Khan University (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: OPP1131320
Record Dates: First submitted 2017-03-08; First posted 2017-07-05 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Malnutrition; Pneumonia; Diarrhea; Sepsis; Bacteremia; HIV/AIDS; TB; Enteropathy; Antibiotic Resistant Strain
Keywords: Malnutrition; Hospitalization; Acute Illness; Pediatric; Post-discharge mortality; Mortality; Cohort; Nested case control; Antimicrobial resistance; Antibiotic; Feeding; Undernutrition
MeSH Terms: conditions — Malnutrition; Pneumonia; Diarrhea; Sepsis; Bacteremia; Acquired Immunodeficiency Syndrome; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, rectal swabs, faeces, urine, peripheral blood mononuclear cells, bacterial isolates, PBMCs, TLR-stimulated whole blood, urine, breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hospitalized children with severe wasting or kwashiorkor (SWK): Children recruited at admission to hospital and followed up for 180 days post-discharge.
- Community reference participants (CP): Children recruited from the community who are seen a single appointment in the community.
- Hospitalized children with moderate wasting (MW): Children recruited at admission to hospital and followed up for 180 days post-discharge.
- Hospitalized children without wasting (NW): Children recruited at admission to hospital and followed up for 180 days post-discharge.

SUMMARY:
The CHAIN Network aims to identify modifiable biomedical and social factors driving the greatly increased risk of mortality among young undernourished children admitted to hospital with acute illness, as inpatients and after discharge. The study will inform priorities, risks and targeting for multi-faceted interventional trials.

CHAIN is a multi-centre cohort study with a nested case control analysis of stored biological samples. Study sites are located in Africa and South Asia. Children will be recruited at admission to hospital, stratified by nutritional status. Exposures will be assessed at admission, during hospitalisation, at discharge, and at two time points after discharge. The main outcomes of interest are mortality, re-admission to hospital and failure of nutritional recovery up to 180 days after discharge. To determine community health norms, an additional sample of children living in the same communities will be enrolled and assessed at one time point only.

DETAILED DESCRIPTION:
Despite an overall reduction of child mortality in LMICs, acutely-ill undernourished children continue to have a greatly elevated risk of death, both during hospitalisation and following discharge. However, we currently lack robust evidence for their management. Factors underlying the risks of mortality may relate to the acute illness itself, to children's longer term health trajectories, or to the home nutritional and care environment. The ultimate goal of the CHAIN Network is to identify and prioritize actionable intervention targets to reduce mortality among acutely ill undernourished children.

CHAIN's initial aim is to better understand the characteristics that determine increased risk of mortality in this vulnerable population, whether biological (related to infection, immunity and metabolism), nutritional (intake and anthropometry), health system factors (affecting management and discharge) or behavioural (community/caregiver interactions). CHAIN brings clinicians and scientists together from a variety of high-burden settings in Africa and South Asia. CHAIN will establish prospective cohorts of acutely ill young children across different geographies with differing population, social and environmental characteristics (stunted vs. wasting, rural vs. urban and presence of risk factors such as malaria and HIV).

Eight sites will be involved, including three hospitals in Kenya (Kilifi County, Migori County and Mbagathi District), two in Bangladesh (Matlab and the icddr,b Dhaka), and one in each of Uganda (Mulago), Malawi (Queen Elizabeth Community Hospital), Pakistan (Civil Hospital Karachi) and in West Africa (TBA). Site will enroll children at admission to hospital, and assess their clinical, social and economic status at admission, during hospitalisation, at discharge and during follow up for 180 days after discharge. The sites will also enrol children from the community to determine community norms (where ill and undernourished children would be expected to typically recover to). Protocols and procedures will be carefully harmonised across sites.

Children aged 2 months to 2 years admitted to hospital will be considered for inclusion and enrolment stratified by nutritional status. Following informed consent, baseline data of prognostic importance, including demographic and social information, a detailed clinical examination, anthropometry and measurement of vital signs, including pulse oximetry, will be collected using a standard proforma. A research blood sample will be collected together with the routine clinical blood draw to minimize the patient's discomfort. Rectal swabs and faecal sample will also be obtained from all children.

During admission, care will be provided according to WHO and national guidelines. Children will be reviewed daily and clinical features, progress and treatment received recorded on a structured case report form. In the event of death in hospital, a standard audit questionnaire will be completed. During admission, primary caregivers, usually the mother, will be interviewed screened for mental health problems. At discharge, anthropometry, a clinical assessment and blood, rectal swab and whole stool collected. Families will be linked with chronic care services where needed.

A home visit will be conducted for all participants, the GPS location recorded. Information homestead infrastructure, water and sanitation, population, livelihood, child care and socioeconomic characteristics. Children will be followed up at 45, 90 and 180 days after discharge. A health questionnaire will document health and social events, and dietary intake. Anthropometry, and faecal and blood samples collected.

Caregivers will be asked to attend the study hospital should the caregiver believes they may require hospitalisation. Study participants who are re-admitted to hospital will undergo standardised clinical assessment including history, examination and sample collection. In the event of death occurring outside the study hospital, a standard verbal autopsy (VA) will be completed by trained staff within 28 days of becoming aware of a death. VAs along with all available information will be used to ascribe causes of death.

Community participants will be invited to the study clinic for assessment. Following informed consent, they will have a clinical examination, anthropometry, blood and stool samples as children who are admitted. Children requiring non-urgent medical care will be eligible for inclusion as community participants but will be given basic treatment in the study clinic and/or referred to appropriate treatment centres. Study staff will refer community participants with incomplete vaccination or requiring care for chronic conditions as needed.

Several domains of exposure will be assessed: demographic, nutrition and metabolism; acute and chronic conditions; community-acquired and nosocomial infections (including antimicrobial resistance); gut function & dysbiosis; inflammation; responses to treatment; and the home care environment.

Successful design of an intervention package to address post-discharge child mortality will require attention social and economic agency and vulnerability, access and interactions with health services, and ethical considerations. A qualitative sub-study will examine these factors in context in rural and urban sites in Kenya and Bangladesh to identify critical social limitations and potential approaches to intervention. These data will inform the network's development, piloting, and implementation of interventions.

Additional sub-studies at a subset of sites will also examine in more detail the diagnosis and role of TB; and changes in functional immune responses; body composition and neurodevelopment during follow up.

ELIGIBILITY:
Inclusion criteria (hospitalized participants):

* Children 2 months-23 months.
* Admitted to hospital.
* Planning to remain within the hospital catchment area and willing to come for specified visits during the 6 month follow up period.
* Parent or guardian consents on child's behalf.

Inclusion criteria (community participants):

* Aged 2 to 23 months
* Living in the same community as the acutely ill children recruited.
* Not having an acute illness requiring hospital admission
* Absence of known, but untreated HIV or TB
* Not admitted to hospital within the last 14 days
* Not previously included in the study
* Parent or guardian consents on child's behalf.

Exclusion Criteria (all participants):

* Requiring immediate resuscitation at admission to hospital*
* Unable to tolerate oral feeds while in his/her usual state of health
* Underlying terminal illness that in the opinion of the treating physician is likely to lead to death within 6 months (e.g., cancer, congenital heart disease)
* Diagnosed with a condition that in the opinion of the treating physician is likely to require surgery within 6 months
* Diagnosed chromosomal abnormality (syndromically or genetically diagnosed abnormality)
* Primary reason for admission is poisoning, trauma or a surgical condition
* Previously enrolled in this study
* Sibling currently or previously enrolled in this study

(* children requiring resuscitation will be defined as those with on-going cardiac or pulmonary arrest or judged to be peri-arrest by the attending physician)

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospital and post-discharge cohort: Children being admitted to hospital.
  Community reference participants: Children living in the same communities as those recruited into the hospitalized cohort.
Sampling Method: Non-Probability Sample
Enrollment: 4335 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 30 days after admission to hospital
  Assessed using clinical and civil records and verbal autopsy
Mortality | Up to 180 days after discharge from hospital
  Assessed using clinical and civil records and verbal autopsy

SECONDARY OUTCOMES:
Rehospitalization | Up to 180 days after discharge from hospital
  Number of participants, assessed from direct observation or clinical records
Change in weight-for-height z-score | Up to 180 days after discharge from hospital
  Post-discharge growth
Change in length-for-age z-score | Up to 180 days after discharge from hospital
  Post-discharge growth
Change in mid-upper arm circumference | Up to 180 days after discharge from hospital
  Post-discharge growth

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkley, MBBS, FRCPCH, Principal Investigator — University of Oxford; Judd L Wilson, MD, MPH, Principal Investigator — University of Washington
Locations (8):
- Bangladesh (2):
  - Matlab Hospital, Dhaka, Chittagong
  - ICDDR,B Dhaka Hospital, Dhaka
- Kenya (3):
  - Kilifi County Hospital, Kilifi
  - Migori County Hospital, Migori
  - Mbagathi District Hospital, Nairobi
- Queen Elizabeth Central Hospital, Blantyre, Malawi
- Civil Hospital Karachi, Karachi, Pakistan
- Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Njunge JM, Tickell K, Diallo AH, Sayeem Bin Shahid ASM, Gazi MA, Saleem A, Kazi Z, Ali S, Tigoi C, Mupere E, Lancioni CL, Yoshioka E, Chisti MJ, Mburu M, Ngari M, Ngao N, Gichuki B, Omer E, Gumbi W, Singa B, Bandsma R, Ahmed T, Voskuijl W, Williams TN, Macharia A, Makale J, Mitchel A, Williams J, Gogain J, Janjic N, Mandal R, Wishart DS, Wu H, Xia L, Routledge M, Gong YY, Espinosa C, Aghaeepour N, Liu J, Houpt E, Lawley TD, Browne H, Shao Y, Rwigi D, Kariuki K, Kaburu T, Uhlig HH, Gartner L, Jones K, Koulman A, Walson J, Berkley J. The Childhood Acute Illness and Nutrition (CHAIN) network nested case-cohort study protocol: a multi-omics approach to understanding mortality among children in sub-Saharan Africa and South Asia. Gates Open Res. 2022 Nov 3;6:77. doi: 10.12688/gatesopenres.13635.2. eCollection 2022. PMID 36415883
- [Derived] Tickell KD, Denno DM, Saleem A, Ali A, Kazi Z, Singa BO, Otieno C, Mutinda C, Ochuodho V, Richardson BA, Asbjornsdottir KH, Hawes SE, Berkley JA, Walson JL. Enteric Permeability, Systemic Inflammation, and Post-Discharge Growth Among a Cohort of Hospitalized Children in Kenya and Pakistan. J Pediatr Gastroenterol Nutr. 2022 Dec 1;75(6):768-774. doi: 10.1097/MPG.0000000000003619. Epub 2022 Sep 20. PMID 36123771
- [Derived] Childhood Acute Illness and Nutrition Network. Childhood Acute Illness and Nutrition (CHAIN) Network: a protocol for a multi-site prospective cohort study to identify modifiable risk factors for mortality among acutely ill children in Africa and Asia. BMJ Open. 2019 May 5;9(5):e028454. doi: 10.1136/bmjopen-2018-028454. PMID 31061058
- See also: The CHAIN Network — http://www.chainnetwork.org/
- See also: Childhood Acute Illness and Nutrition (CHAIN) Network: a protocol for a multi-site prospective cohort study to identify modifiable risk factors for mortality among acutely ill children in Africa and Asia — https://bmjopen.bmj.com/content/9/5/e028454.long